CLINICAL TRIAL: NCT02760732
Title: Drug Eluting Balloon Combined With Cutting Balloon for Treatment of Unstable Angina
Brief Title: Drug Eluting Balloon for Treatment of Unstable Angina
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yun Dai Chen (Other)
Responsible Party: Sponsor-Investigator, Yun Dai Chen, MD, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301_xnk1
Record Dates: First submitted 2016-02-29; First posted 2016-05-04 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Angina, Unstable
MeSH Terms: conditions — Angina, Unstable | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- drug eluting balloon group (Experimental): patients with unstable angina were randomised to drug eluting balloon group for percutaneous transluminal coronary angioplasty with a strategy of cutting balloon(Flextome Cutting Balloon, Boston Scientific Corporation, US) pre-dilation first and then drug eluting balloon(Sequent please; B. Braun, Melsungen, Germany) .
  Interventions: Device: drug eluting balloon; cutting balloon
- drug eluting stent group (Experimental): patients with unstable angina were randomised to this group for drug eluting stent (YINYI® Polymer-free Drug-coated (Paclitaxel) Coronary Stent System, Liaoning Biomedical Materials R&D Center Co., Ltd. China) implantation.
  Interventions: Device: drug eluting stent

INTERVENTIONS:
Device: drug eluting balloon; cutting balloon — Patients eligible for inclusion criteria were randomised to study group for percutaneous transluminal coronary angioplasty with a strategy of cutting balloon pre-dilation first and then drug eluting balloon.
  Other Names: Sequent please; B. Braun; Flextome Cutting Balloon, Boston Scientific
  Arms: drug eluting balloon group
Device: drug eluting stent — with a strategy of drug-eluting stent implantation alone for de novo coronary artery lesions.
  Other Names: YINYI®
  Arms: drug eluting stent group

SUMMARY:
This study was to investigate the effect and safety of drug eluting balloon combined for treatment of unstable angina.

DETAILED DESCRIPTION:
Patients with unstable angina were randomized to drug eluting stent only or drug eluting balloon group. Angiographic follow-up was performed after 12 months. The primary endpoints were late lumen loss (LLL) and the secondary endpoints were target lesion revascularization (TLR),and the major adverse cardiovascular events (MACE) .

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18, < 80 years old, with unstable angina
* Single-vessel or double-vessel disease
* Length of target lesion < 25mm
* Diameter of target vessel >2.5mm, < 3.5mm

Exclusion Criteria:

* Left main disease
* Chronic total occlusion
* Severe Tortuosity
* Heavy calcification
* Severe liver failure, moderate or severe kidney failure
* Malignant disease
* Active infectious disease
* Pregnancy or breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-06-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Target Lumen assessed by optical coherence tomography | 12 months
  A coronary de novo lesion in patient after intervened was measured with optical coherence tomography .To measure the changes in target lumen at 12 months.

SECONDARY OUTCOMES:
Incidence rate of MACE | Incidence rate of MACE from baseline to 12 months
  MACE include composite of death, myocardial infarction, or target-vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: CHEN YUN DAI, MD, Principal Investigator — The General Hospital of PLA
Locations (1):
- The General Hospital of PLA, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li B, Ding Y, Tian F, Chen W, Han T, Chen Y. Assessment of a Drug-Eluting Balloon for the Treatment of de novo Coronary Lesions Guided by Optical Coherence Tomography: Study Protocol for a Randomized Controlled Trial. Cardiology. 2017;136(4):252-257. doi: 10.1159/000452125. Epub 2016 Nov 16. PMID 27846629